CLINICAL TRIAL: NCT03726996
Title: Novel Off-label Use of Desipramine in Infantile Neuroaxonal Dystrophy: Targeting the Sphingolipid Metabolism Pathway to Reduce Accumulation of Ceramide.
Brief Title: Desipramine in Infantile Neuroaxonal Dystrophy (INAD).
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding exhausted
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100799
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-08

CONDITIONS: Infantile Neuroaxonal Dystrophy
Keywords: Pediatric genetic disorder; cognitive function; neuro-muscular disorder; PLA2G6
MeSH Terms: conditions — Neuroaxonal Dystrophies | interventions — Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with INAD (Experimental): Infantile neuroaxonal dystrophy (INAD) is an extremely rare autosomal recessive neurodegenerative disorder that has grave clinical outcome and significant morbidity and mortality.
  Interventions: Drug: Desipramine

INTERVENTIONS:
Drug: Desipramine — Study drug (desipramine) provided in tablet form to be taken daily.

SUMMARY:
This is a research study to find out if clinically prescribed desipramine is effective at improving the symptoms and slowing the progression of Infantile Neuroaxonal Dystrophy (INAD) in affected children.

Participants will receive an initial oral dose of study drug once a day. This dose may be changed depending on response to study drug Clinically collected data will be recorded for up to 5 years. Investigators will also ask for participant permission to obtain a sample of child's skin biopsy from unused clinical sample previously collected for standard of care.

DETAILED DESCRIPTION:
To be eligible participants must be able to swallow tablets The study drug is to be taken once daily Schedule of events. Day 0 - ECG and blood tests (4 ml or ¾ teaspoon) Day 3 - ECG and blood tests (4 ml or ¾ teaspoon) Day 7 - ECG and blood tests (4 ml or ¾ teaspoon) Weeks 2, 3, 4, 8 & 12. ECG and blood tests (4 ml or ¾ teaspoon) Every 3 months for up to 5 years.

.

ELIGIBILITY:
Inclusion Criteria:

* 03-17years.
* Any gender
* Confirmed homozygotes or compound heterozygotes of pathogenic mutation variant(s) in PLA2G6
* Confirmed homozygotes of pathogenic mutation in PLA2G6
* Documentation of clinical presentation (signs and symptoms of neurodegenerative process) of INAD

Exclusion Criteria:

* Patient has sign and symptom suggesting an ongoing acute or chronic illness such as fever of unknown origin or infection.
* Patient has a second genetic condition
* Parents are unable or unwilling to return for continued care for up to 12 months

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong-hui Jiang, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Children With INAD
Started | 4
Completed | 0
Not Completed | 4
Not completed — Parent's decision | 2
Not completed — Study early termination | 2

BASELINE CHARACTERISTICS:
Arm/Group | Children With INAD
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
Gross Motor Function Measure (GMFM-66) [Number; unit: units on a scale] — The GMFM-66 is a 66 item standardized observational instrument used to measure change in gross motor function over time in children. A unit of change has the same meaning throughout the scale ranging from 0 to 100. 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Scoring the GMFM-66 requires the use of a computer program called the Gross Motor Ability Estimator (GMAE). Individual item scores are entered and a mathematical algorithm calculates an interval level total score. The total score is an estimate of the child's gross motor function. Population: Data collected on one participant.
  units on a scale
    number analyzed (Participants) | 1
    (all) | 1
Quick Motor Function Test (QMFT) [Number; unit: units on a scale] — The QMFT is a 16 item psychometrically robust outcome assessment validated in children and adults with Pompe disease (a lysosomal storage disorder characterized by progressive muscle weakness). This motor function test observes performance and scores the items separately on a 5-point ordinal scale (ranging from 0 to 4). If items can be performed on both left and right extremities, the right side is taken. A total score is obtained by adding the scores of all items. The total score ranges between 0 and 64 points. A higher score correlates with greater motor function. Population: Data collected on one participant.
  units on a scale
    number analyzed (Participants) | 1
    (all) | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Gross Motor Function as Measured by Gross Motor Function Measure (GMFM-66)
Description: The Gross Motor Function Measure (GMFM-66) is a 66 item standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. Items are ordered in terms of difficulty and a unit of change has the same meaning throughout the scale ranging from 0 to 100. 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Scoring the GMFM-66 requires the use of a computer program called the Gross Motor Ability Estimator (GMAE). Individual item scores are entered and a mathematical algorithm calculates an interval level total score. The total score is an estimate of the child's gross motor function.
Time Frame: Baseline, 3, 6, 9, and 12 months
Population: No data collected beyond baseline.
Arm/Group | Children With INAD
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Motor Function as Measured by Quick Motor Function Test (QMFT)
Description: The Quick Motor Function Test (QMFT) is a 16 item, psychometrically robust outcome assessment, validated in children and adults with Pompe disease (a lysosomal storage disorder characterized by progressive muscle weakness). This motor function test observes performance and scores the items separately on a 5-point ordinal scale (ranging from 0 to 4). If items can be performed on both left and right extremities, the right side is taken. A total score is obtained by adding the scores of all items. The total score ranges between 0 and 64 points. A higher score correlates with greater motor function.
Time Frame: Baseline, 3, 6, 9, and 12 months
Population: No data collected beyond baseline.
Arm/Group | Children With INAD
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Cognitive Function as Measured by the Vineland Adaptive Behavioral Scale
Description: The Vineland-3 is a standardized measure of adaptive behavior--the things that people do to function in their everyday lives. It is a norm-based instrument that compares the examinee's adaptive functioning in four domains: Communication, Daily Living Skills, Socialization and Motor Skills to that of others of the same age. A composite score of adaptive behavior is calculated that summarizes the individual's performance across all four domains.
Time Frame: Baseline, 3, 6, 9, and 12 months
Population: Data not collected.
Arm/Group | Children With INAD
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Participants With Change in Q-T Interval on ECG
Description: Evidence of ECG changes, specifically, prolonged Q-T interval in response to study drug. The Q-T interval is the time from the start of the Q wave to the end of the T wave. It represents the time taken for ventricular depolarisation and repolarisation, effectively the period of ventricular systole from ventricular isovolumetric contraction to isovolumetric relaxation. Participants with a prolonged Q-T interval at any timepoint is reported.
Time Frame: Baseline, 3, 6, 9, and 12 months
Population: No data collected beyond 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With INAD
Number analyzed (Participants) | 4
Participants | 1

5. Primary Outcome: Number of Participants With Abnormal Transaminase Values
Description: Transaminase values as measured by serum alanine transaminase (ALT) and aspartate transaminase (AST). Participants with abnormal transaminase values at any timepoint is reported.
Time Frame: Baseline, 3, 6, 9, and 12 months
Population: No data collected beyond 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With INAD
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 7 months
Description: ECG and safety lab prior to initial dose, at days 3 & 7 post initial dose and after each dose change. PI assessment no less frequently than every 12 weeks.
Arm/Group | Children With INAD
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Early termination due to relocation of PI from our clinical study site. All assessments were halted before the end of the study. Insufficient data collected to draw any conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT03726996/Prot_SAP_000.pdf